CLINICAL TRIAL: NCT06933537
Title: This Study is Designed to Evaluate the Efficacy of Personalized Alternating Current Stimulation in the Treatment of Emotional Disorders in Patients With Inflammatory Demyelination of the Central Nervous System
Brief Title: Effectiveness of Personalized Alternating Current Stimulation for Treating Emotional Disorders in CNS Demyelination Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: xw-tES-02
Record Dates: First submitted 2025-01-19; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Idiopathic Inflammatory Demyelinating Disorders of the Central Nervous System

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neuromodulation Group (Active Comparator)
  Interventions: Device: Neuroelectrics StarStim 32
- Sham-Neuromodulation Group (Sham Comparator)
  Interventions: Device: Neuroelectrics StarStim 32

INTERVENTIONS:
Device: Neuroelectrics StarStim 32 — Using the advanced Neuroelectrics StarStim 32 device from Spain, individualized imaging modeling systems are employed to precisely target the frontal cortex. Personalized EEG-guided electrical stimulation protocols are selected. The stimulation parameters are as follows: a current intensity of 2 mA, a duration of 21 minutes per session, once daily for five consecutive days, with EEG monitoring conducted before and after electrical stimulation.
  Arms: Neuromodulation Group
Device: Neuroelectrics StarStim 32 — Sham stimulation is performed using the same device and procedures as the neuromodulation group. The stimulator automatically shuts off after 30 seconds, while maintaining the device's connection. This design creates an initial sensation similar to actual stimulation while preserving the double-blind nature of the study.
  Arms: Sham-Neuromodulation Group

SUMMARY:
This study is designed to evaluate the efficacy of personalized alternating current stimulation in the treatment of emotional disorders in patients with inflammatory demyelination of the central nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with inflammatory demyelinating diseases of the central nervous system, such as neuromyelitis optica spectrum disorders (NMOSD) and multiple sclerosis (MS)
* Hamilton Anxiety Scale (HAM-A) score > 14
* Aged between 18 and 65 years, with no gender restrictions
* Receiving stable doses of immunosuppressive therapy for at least one month
* Expanded Disability Status Scale (EDSS) score ≤ 6
* Right-handed
* Willing to participate and sign informed consent

Exclusion Criteria:

* Recorded relapse within the past month
* Recent medication adjustments or treatments involving modified electroconvulsive therapy, transcranial magnetic stimulation, or other neuromodulation techniques within the past month
* Participation in any other clinical study within the past month or currently
* Presence of cochlear implants, cardiac pacemakers, or implanted stimulators in the brain
* Impaired skin integrity at the electrode placement site or allergies to electrode gel or adhesives
* History of epilepsy, hydrocephalus, central nervous system tumors, brain injury, or intracranial infections
* Pregnant or breastfeeding women, or those planning to conceive in the near future
* Hamilton Depression Scale suicide item score ≥ 3 or comorbid severe mental disorders
* Presence of severe or unstable organic diseases
* Poor compliance preventing cooperation with treatment, follow-up, or clinical, EEG, and imaging data collection
* Any condition deemed unsuitable for study participation by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-12-29 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
HAMA (Hamilton Anxiety Rating Scale) | From enrollment to the end of treatment at 1month
  A clinician-administered scale used to assess the severity of a patient's anxiety based on a series of symptoms.
  Range: 0-56
  Higher Scores: Indicate more severe anxiety.
  Purpose: Used to evaluate the severity of anxiety symptoms in patients, primarily in clinical and research settings.
HADS (Hospital Anxiety and Depression Scale) | From enrollment to the end of treatment at 1month
  Description:
  A self-report scale used to identify the levels of anxiety and depression in patients, particularly in a hospital setting. It consists of 14 items, split into two subscales: one for anxiety and one for depression.
  Range: 0-42 (for each subscale)
  Higher Scores: Indicate higher levels of anxiety or depression.
  Purpose: Used for screening and evaluating the severity of anxiety and depression in patients, especially those with physical illnesses.
SPS (Social Phobia Scale) | From enrollment to the end of treatment at 1month
  A self-report scale used to measure the severity of social anxiety or social phobia.
  Range: 0-120
  Higher Scores: Indicate greater severity of social anxiety.
  Purpose: Used to assess the intensity of social anxiety and its impact on the individual's daily life.
PSWQ (Penn State Worry Questionnaire) | From enrollment to the end of treatment at 1month
  A self-report scale used to assess the frequency and intensity of a person's worry.
  Range: 16-80
  Higher Scores: Indicate more frequent and intense worry.
  Purpose: Primarily used in research and clinical settings to evaluate generalized anxiety and worry tendencies.

SECONDARY OUTCOMES:
EDSS (Expanded Disability Status Scale) | From enrollment to 1 month later
  A clinician-administered scale used to measure the severity of disability in patients with multiple sclerosis (MS). It assesses neurological impairment in eight functional systems.
  Range: 0-10
  Higher Scores: Indicate greater disability, with 0 representing normal neurological function and 10 representing death due to MS.
  Purpose: Used to assess the degree of disability and monitor changes over time in MS patients.
FSS (Fatigue Severity Scale) | From enrollment to 1 month later
  A self-report scale designed to assess the impact of fatigue on a patient's daily life. It evaluates the intensity of fatigue in relation to physical activities, work, and social life.
  Range: 9-63
  Higher Scores: Indicate more severe fatigue.
  Purpose: Used primarily in multiple sclerosis and other neurological disorders to quantify fatigue severity.
HAMD (Hamilton Depression Rating Scale) | From enrollment to 1 month later
  A clinician-administered scale used to assess the severity of depression in patients, based on mood, feelings of guilt, and somatic symptoms.
  Range: 0-52
  Higher Scores: Indicate more severe depression.
  Purpose: Primarily used to assess depression severity in clinical settings and for treatment evaluation.
MMSE (Mini-Mental State Examination) | From enrollment to 1 month later
  A brief 30-point test used to screen for cognitive impairment and assess the level of cognitive function in patients, focusing on orientation, memory, and attention.
  Range: 0-30
  Higher Scores: Indicate better cognitive function, with scores below 24 suggesting cognitive impairment.
  Purpose: Used to assess cognitive function, often in patients with suspected dementia or other cognitive disorders.
MoCA (Montreal Cognitive Assessment) | From enrollment to 1 month later
  A screening tool used to detect mild cognitive impairment. It evaluates multiple cognitive domains, including attention, memory, language, and executive function.
  Range: 0-30
  Higher Scores: Indicate better cognitive function, with a score below 26 typically suggesting cognitive impairment.
  Purpose: Commonly used to assess cognitive function in patients with early dementia, stroke, or neurological disorders.
SDMT (Symbol Digit Modalities Test) | From enrollment to 1 month later
  A neuropsychological test assessing processing speed, attention, and visual-motor coordination. It requires the patient to match symbols to digits based on a key.
  Range: Varies based on time and performance (measured in seconds or correct responses).
  Higher Scores: Indicate better processing speed and cognitive function.
  Purpose: Used to assess cognitive performance and processing speed in clinical research and patient assessments.
DST (DigiScan Test) | From enrollment to 1 month later
  A neuropsychological test used to evaluate attention and working memory by requiring patients to process and manipulate digital sequences.
  Range: Dependent on the version of the test used (typically time-based or score-based).
  Higher Scores: Indicate better cognitive performance, particularly in attention and working memory.
  Purpose: Assesses cognitive function, often used in the evaluation of neurodegenerative diseases or brain injury.
BVMT (Brief Visuospatial Memory Test) | From enrollment to 1 month later
  A test designed to measure visuospatial memory and learning ability, asking patients to remember and recall spatially presented objects.
  Range: Varies depending on the test format (measured in correct responses or recall time).
  Higher Scores: Indicate better visuospatial memory performance.
  Purpose: Used to assess memory, particularly in the context of cognitive disorders like MS and Alzheimer's disease.
NRS (Numerical Rating Scale) | From enrollment to 1 month later
  A self-reported scale that asks patients to rate the intensity of their pain on a scale from 0 to 10.
  Range: 0-10
  Higher Scores: Indicate more intense pain.
  Purpose: Commonly used in clinical practice to measure pain intensity and assess treatment efficacy.
SF-MPQ (Short-Form McGill Pain Questionnaire) | From enrollment to 1 month later
  A self-reported questionnaire used to assess the quality and intensity of pain, measuring sensory, affective, and evaluative dimensions of pain.
  Range: 0-78 (higher scores indicate greater pain severity)
  Higher Scores: Indicate greater pain intensity and distress.
  Purpose: Often used to assess pain in clinical and research settings, providing both quantitative and qualitative measures of pain.
ESS (Epworth Sleepiness Scale) | From enrollment to 1 month later
  A self-report questionnaire used to assess daytime sleepiness and the likelihood of falling asleep in various situations.
  Range: 0-24
  Higher Scores: Indicate higher levels of daytime sleepiness.
  Purpose: Used to assess sleepiness, often in the context of sleep disorders like sleep apnea or narcolepsy.
Ashworth Scale | From enrollment to 1 month later
  A clinician-administered scale used to measure muscle spasticity. It evaluates the resistance of a muscle to passive movement in response to varying speeds.
  Range: 0-4
  Higher Scores: Indicate greater spasticity, with 0 being no spasticity and 4 being severe spasticity.
  Purpose: Commonly used in neurological conditions such as cerebral palsy, multiple sclerosis, and stroke.
SF-36 (Short Form 36 Health Survey) | From enrollment to 1 month later
  A self-reported health survey designed to measure quality of life, including physical, emotional, and social well-being. It consists of 36 questions grouped into eight domains.
  Range: 0-100 for each domain (higher scores indicate better health status).
  Higher Scores: Indicate better health and quality of life.
  Purpose: Used widely to assess general health status, particularly in chronic illness and clinical trials.
CGI-I (Clinical Global Impression - Improvement) | From enrollment to 1 month later
  A clinician-administered scale that evaluates the overall improvement of a patient's condition since the initiation of treatment.
  Range: 1-7
  Higher Scores: Indicate less improvement, with a score of 1 indicating "very much improved" and 7 indicating "very much worse."
  Purpose: Used to assess treatment effectiveness in clinical trials and practice, particularly in psychiatric and neurological conditions.
EGI Recording EEG Data and MRI Data | From enrollment to 1 month later
  EEG (Electroencephalography): A technique used to measure electrical activity in the brain. It records brain waves and can help identify abnormalities related to seizures, sleep disorders, or other neurological conditions.
  MRI (Magnetic Resonance Imaging): A non-invasive imaging technique that uses magnetic fields and radio waves to create detailed images of organs and tissues. It is commonly used to assess brain structure, identify lesions, and detect abnormalities.
  Purpose: Both EEG and MRI are used to monitor and assess brain activity and structure in patients, providing valuable insights into neurological conditions and helping in diagnosis and treatment planning.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No